CLINICAL TRIAL: NCT06873178
Title: Liver Metastasis of Pancreatic Cancer：Chinese Surgical Study Group
Brief Title: The Significance and Indications of Surgery for Synchronous Liver Metastatic Pancreatic Cancer
Acronym: PCLM:CSSG
Status: Active, not recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Peking University First Hospital (Other); Chongqing General Hospital (Other); Tongji Hospital (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Zhiying Yang, Director, Head of Hepatobiliary and Pancreatic Surgery, Clinical Professor, China-Japan Friendship Hospital
Other Study IDs: 2024-KY-385-2; MR-11-25-016581 (Other: National Health Security Information Platform Medical Research Registration and Filing Information System)
Record Dates: First submitted 2025-03-02; First posted 2025-03-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer; Liver Metastases; Surgery; Adjuvant Therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- retrospective: Retrospectively collect cases of pancreatic cancer with synchronous liver metastasis treated and analyze the preliminary results.
- foresight: On the basis of retrospective studies, a prospective clinical study is conducted. Through the prospective study of the outcomes of systemic treatment for patients with pancreatic cancer liver metastasis and the clinical results of surgical treatment after the effectiveness of systemic treatment, a basis is provided for the diagnosis and treatment strategies of pancreatic cancer liver metastasis.

SUMMARY:
To explore the clinical characteristics of pancreatic cancer patients with liver metastases who can benefit from surgery, and to develop evaluation criteria for surgical indications, so as to provide basis for comprehensive treatment strategies for advanced pancreatic cancer patients.

DETAILED DESCRIPTION:
Initial Systemic Treatment: Subjects who meet the inclusion criteria will first undergo systemic treatment. The primary treatment regimens will follow the NCCN guideline-recommended first-line chemotherapy options, including the AG regimen, FOLFIRINOX regimen, and the NALIRIFOX regimen.

Periodic Assessments: Every 4 treatment cycles, laboratory tests (including blood routine, coagulation function, liver and kidney function, and tumor markers) and imaging studies (enhanced CT or MRI, with PET-CT if necessary) will be conducted. After 4-6 cycles, imaging and tumor marker assessments will be performed to evaluate the patient's disease status. A multidisciplinary discussion will determine if patients with a good response to systemic treatment are eligible for radical surgery.

Treatment Adjustment and Surgical Intervention: For patients assessed as having disease progression during the first evaluation, the treatment plan will be adjusted, and assessments will be conducted every 2 cycles. Patients showing a good response may still be considered for radical surgery. For pancreatic lesions, surgical procedures such as pancreaticoduodenectomy or distal pancreatectomy with splenectomy will be performed based on the lesion's location, with total pancreatectomy considered if necessary. For liver lesions, the surgical approach will depend on the number, size, and location of the lesions. During surgery, tumor and adjacent tissue samples (approximately 100mg, the size of a soybean) will be collected for research purposes, provided it does not affect diagnosis. Postoperative discarded specimens (approximately 500mg) will also be collected and preserved.

Postoperative Monitoring: Laboratory tests, including but not limited to blood routine, coagulation, liver, kidney, and pancreatic function, will be collected on postoperative days 1, 3, 5, 7, and 30.

Adjuvant Treatment and Complication Monitoring: Postoperative adjuvant treatment will continue according to the original regimen. Any postoperative complications and adverse reactions during chemotherapy will be recorded.

Trial Progress Tracking: The progress of each subject will be documented. If a subject withdraws or drops out, the reason and the date of the last medication will be recorded.

Follow-Up: After the completion of treatment, patients will be followed up monthly until death.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* Pancreatic cancer was diagnosed as pancreatic ductal adenocarcinoma by biopsy of primary/metastases
* Physical Condition Score (ECOG)0-1
* Simultaneous/prior discovery of liver metastases and primary lesions was defined as simultaneous liver metastases
* Enhanced CT/MRI can detect liver metastases (if the diseases not detected by enhanced CT/MRI during screening are not included in the number calculation)
* The patient's liver, kidney and bone marrow function is good

Exclusion Criteria:

* The primary lesions of pancreatic cancer are acinar cell carcinoma of pancreas, neuroendocrine carcinoma of pancreas and other pathological types
* there are other metastases outside the liver
* Had other malignant tumors within 5 years
* History of central nervous system disease, mental illness, unstable angina pectoris, congestive heart failure, severe arrhythmia and other serious diseases
* Active or chronic hepatitis B/C virus infection
* Allergy to iodine, unable to perform enhanced imaging
* Previous anti-tumor therapy for pancreatic cancer (surgery/ radiotherapy/ chemotherapy/ ablation/ targeted therapy/ immunotherapy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
OS | through study completion, an average of 2 year
  Overall Survival

SECONDARY OUTCOMES:
RFS | through study completion, an average of 2 year
  Recurrence free survival

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China